CLINICAL TRIAL: NCT03477318
Title: Accuracy of Endoscopists in Predicting Polyp Pathology
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 17-075
Record Dates: First submitted 2018-03-20; First posted 2018-03-26 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2018-05

CONDITIONS: Resected Polyp
Keywords: colonoscopy, polyp, endoscopist
MeSH Terms: conditions — Polyps

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing screening colonoscopy: Patients undergoing first-time colonoscopy using white light with at least 1 polyp resected.

SUMMARY:
The study purpose is to assess the accuracy of experienced endoscopists at a community hospital in predicting histological types of polyps resected at colonoscopy using white light. Patients 50 years or older undergoing first-time screening colonoscopy will be included in this observational study.

DETAILED DESCRIPTION:
The study purpose is to assess the accuracy of experienced endoscopists at a community hospital in predicting histological types of polyps resected at colonoscopy using white light. The study will be conducted at Good Samaritan Hospital and TriHealth Surgery Center West. Study participants include patients 50 years or older undergoing first-time screening colonoscopy. This is an observational study and does not involve any patient interventions. After completing the colonoscopy, the endoscopist will document their prediction of the polyp type. The polyp type predicted by the endoscopist will be compared to the polyp type documented in the pathology report to determine accuracy. It is estimated that study enrollment will take 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Males and females

Exclusion Criteria:

* first degree relative diagnosed with colorectal carcinoma at age 59 or under
* New onset of iron deficiency anemia (within past 3 months)
* Abnormal imaging of colon within past 3 months
* Pregnant women
* Inadequate visualization reported by endoscopist

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients 50 years or older undergoing first-time screening colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2018-11-07 (Actual)

PRIMARY OUTCOMES:
Polyp prediction accuracy | up to 5 days
  Accuracy of predicting polyp type

CONTACTS AND LOCATIONS:
Locations (1):
- Good Samaritan Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No